CLINICAL TRIAL: NCT07095504
Title: Destination Cardiac Rehab: A Multicenter Feasibility Clinical Trial of an Enhanced Virtual World-based Cardiac Rehabilitation Intervention to Improve Cardiovascular Health and Outcomes Among Cardiac Patients
Brief Title: A Study of Cardiac Rehabilitation Intervention to Improve Cardiovascular Health and Outcomes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, LaPrincess C. Brewer, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 25-002186
Record Dates: First submitted 2025-07-24; First posted 2025-07-31 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Cardiovascular Health

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Subject enrolled in a cardiac rehab program (Experimental)
  Interventions: Behavioral: Virtual World-based Cardiac Rehabilitation (VWCR) program

INTERVENTIONS:
Behavioral: Virtual World-based Cardiac Rehabilitation (VWCR) program — 36 Virtual World-based Cardiac Rehabilitation sessions over the course of 12 weeks (3 sessions/week)

SUMMARY:
A single-group, multi-center, non-randomized clinical trial will be conducted to assess the feasibility of implementing an enhanced virtual world-based cardiac rehabilitation (VWCR) program within a muti-site clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Indication for CR according to Centers for Medicare & Medicaid Services (CMS) guidelines (diagnosed within the preceding 12 months) to include one or more of the following:

  * Myocardial infarction
  * Coronary artery bypass surgery
  * Current stable angina (chest pain)
  * Heart valve repair or replacement
  * Percutaneous transluminal coronary angioplasty (PTCA) or coronary stenting
  * Heart or heart-lung transplant
  * Stable chronic heart failure
* Receiving care at one of the participating CR centers
* Age ≥18 years
* Basic Internet navigation skills
* Active email address
* Access to Internet at home or public access (church, library, etc) for 3 virtual visits per week

Exclusion Criteria:

* High risk patients according to the AACVPR risk stratification44 given safety concern of unsupervised exercise

  * Patients receiving continuous inotropic support
  * Recent receipt of a mechanical support device
  * Presence of hemodynamically unstable dysrhythmias (e.g., ventricular tachycardia)
  * Decompensated heart failure
  * Symptomatic valvular heart disease
  * Uncontrolled angina
* Pregnancy (due to associated hormonal and weight changes) per patient report
* Receiving continuous inotropic support
* Presence of a mechanical circulatory support device
* Decompensated heart failure
* Symptomatic valvular heart disease
* Uncontrolled angina
* Presence of hemodynamically unstable dysrhythmias (e.g., ventricular tachycardia) given safety concern of unsupervised exercise
* Visual/hearing impairment or mental disability that would preclude independent use of the VW platform
* Non-English-speaking patients due to logistical challenges with real time translation over a virtual platform
* Currently participating in a cardiac rehab program

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Change in Cardiovascular health score | Baseline, 3 Months, 6 Months
  Cardiovascular health score will be determined by the American Heart Association's (AHA) Life's Simple 8 (LS8). The scale is 0-100 pts (low to high), with LE8 categories as low (0-49), moderate (50-79) and high (80-100). A higher score indicates higher cardiovascular health.
Percent of Virtual world-based cardiac rehabilitation attended | Baseline, 6 Months
  Virtual world-based cardiac rehabilitation attended will be determined by the number of sessions prescribed vs the number of sessions attended (reported as a percent).

SECONDARY OUTCOMES:
Number of cardiovascular hospital readmissions | Baseline, 6 Months
  Cardiovascular Hospital readmissions will be determined by the number of times a patient is admitted to the hospital after initial admission.
All-cause mortality | 6 Months
  All-cause mortality will be determined by the number of patient deaths no matter the cause.

CONTACTS AND LOCATIONS:
Overall Officials: LaPrincess Brewer, M.P.H., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - University of California (UCI), Irvine, Irvine, California
  - Mayo Clinic, Jacksonville, Florida
  - Mayo Clinic, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No